CLINICAL TRIAL: NCT02350465
Title: Detection and Treatment of Sarcopenia and Myosteatosis in Older African Americans
Acronym: ARMS-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E1854-W; MIRB01714 (Other: Washington D.C. Veterans Affairs Medical Center)
Record Dates: First submitted 2015-01-19; First posted 2015-01-29 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Sarcopenia
Keywords: sarcopenia; aging; myosteatosis; exercise; screening
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eccentric Exercise (Experimental): Supervised strengthening exercise using eccentric muscle actions.
  Interventions: Behavioral: Eccentric Exercise
- Concentric Exercise (Active Comparator): Supervised strengthening exercise using concentric muscle actions.
  Interventions: Behavioral: Concentric Exercise

INTERVENTIONS:
Behavioral: Eccentric Exercise — Submaximal progressive resistance exercise (PRE) using eccentric muscle actions for the knee extensors/flexors will be performed for 10 repetitions, 3 to 4 sets, twice per week for 12 weeks.
  Other Names: Negative work training
  Arms: Eccentric Exercise
Behavioral: Concentric Exercise — Submaximal progressive resistance exercise (PRE) using concentric muscle actions for the knee extensors/flexors will be performed for 10 repetitions, 3 to 4 sets, twice per week for 12 weeks.
  Other Names: Conventional strength training
  Arms: Concentric Exercise

SUMMARY:
The objectives of this study are to: 1) validate a rapid, portable, cost-effective method for screening myosteatosis and sarcopenia using diagnostic ultrasound, and 2) investigate a novel approach to progressive resistance exercise involving eccentric muscle actions that will counter the local effects of myosteatosis and sarcopenia in African Americans.

DETAILED DESCRIPTION:
The rationale for this study is the need to proactively address health disparities associated with age-related skeletal muscle dysfunction. Age-related changes in muscle may be characterized by sarcopenia (i.e., loss of muscle mass) and/or myosteatosis (i.e., excessive intramuscular adipose tissue). These changes may result in physical impairments that may be exacerbated by the lack of a formal screening and diagnosis process for older adults in standard healthcare settings. Myosteatosis may compound the effects of sarcopenia and play a significant role the age-related functional decline and higher incidence of type 2 diabetes observed in African Americans in comparison to other ethnic/racial groups. The initial phase of the study will involve the assessment of older African Americans (n = 70) to characterize muscle size and quality in comparison to a younger reference group (n = 70). Participants randomly selected from the older subject pool will be assigned to either the Eccentric Exercise Group or the Concentric Exercise Group for 12 weeks of a supervised strengthening exercise regimen.

ELIGIBILITY:
Inclusion Criteria:

* An African American adult.
* Between 18 and 30 years of age, or between 65 and 85 years of age.
* Able to independently walk at home and in your community (use of an assistive device like a cane or a walker is acceptable).

Exclusion Criteria:

* Uncontrolled hypertension or other cardiovascular disease.
* A Body Mass Index of 32.5 or above may be an exclusion criterion if the X-ray technician determines that dimensions of the scanning bed are not adequate for a reliable examination.
* A musculoskeletal condition that would stop you from performing the physical assessment tests.
* Muscle weakness due to neurological disease or injury (such as stroke or spinal cord injury).
* Moderate to severe sepsis (blood infection) or edema (such as swelling of a limb).
* Been hospitalized over the last three months.
* History of a broken arm or leg bone because of osteoporosis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Sonographic Lean Body Mass at 3 months | At study baseline for all subjects, and at Week 6 and 12 of the intervention period for subjects randomly assigned to an exercise group
  US estimates of aggregate regional LBM (muscle thickness, cm), will be assessed using B-mode diagnostic US with a 13-6 megahertz (MHz) linear array transducer for morphology measures at 6 axial and appendicular sites.

SECONDARY OUTCOMES:
Change from Baseline in dual-energy X-ray absorptiometry (DXA) scanning at 3 months | At study baseline for all subjects, and at Week 12 of the intervention period for subjects randomly assigned to an exercise group
  Participants will undergo DXA scanning in the supine position per manufacturer guidelines to estimate absolute and percentage of total lean body mass (LBM) and body fat (BF).
Change from Baseline in metabolic status at 3 months | At study baseline for all subjects
  A blood sample (60 cc) will be obtained after an 8-hour overnight fast: glucose and insulin levels will be assessed. Other laboratory values will be obtained such as a standard lipid profile and glycated hemoglobin (HbA1C).
Change from Baseline in intramuscular adipose tissue assessment at 3 months | At study baseline for all subjects
  Estimates of intramuscular adipose tissue (IMAT) will be obtained with magnetic resonance imaging using a whole body transmit/receive coil for T2 fat image acquisition of the thigh (dominant side) will be obtained at the mid-femur region.
Change from Baseline in strength assessment at 3 months | At study baseline for all subjects, and at Week 6 and 12 of the intervention period for subjects randomly assigned to an exercise group
  Grip strength will be assessed bilaterally; isometric and isokinetic knee extension/flexion torques will be obtained bilaterally using a dynamometer. Peak concentric torque (at 60 /s and 180 /s) will be obtained in a randomized fashion with subject positioning and stabilization per the manufacturer operations manual.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harris-Love, DSc MPT BS, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (3):
- United States (3):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Howard University, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris-Love MO, Adams B, Hernandez HJ, DiPietro L, Blackman MR. Disparities in the consequences of sarcopenia: implications for African American Veterans. Front Physiol. 2014 Jul 7;5:250. doi: 10.3389/fphys.2014.00250. eCollection 2014. No abstract available. PMID 25071595
- [Background] Harris-Love MO, Monfaredi R, Ismail C, Blackman MR, Cleary K. Quantitative ultrasound: measurement considerations for the assessment of muscular dystrophy and sarcopenia. Front Aging Neurosci. 2014 Jul 14;6:172. doi: 10.3389/fnagi.2014.00172. eCollection 2014. No abstract available. PMID 25071570
- [Background] Harris-Love MO, Seamon BA, Teixeira C, Ismail C. Ultrasound estimates of muscle quality in older adults: reliability and comparison of Photoshop and ImageJ for the grayscale analysis of muscle echogenicity. PeerJ. 2016 Feb 22;4:e1721. doi: 10.7717/peerj.1721. eCollection 2016. PMID 26925339
- [Result] Harris-Love MO, Benson K, Leasure E, Adams B, McIntosh V. The Influence of Upper and Lower Extremity Strength on Performance-Based Sarcopenia Assessment Tests. J Funct Morphol Kinesiol. 2018 Dec;3(4):53. doi: 10.3390/jfmk3040053. Epub 2018 Nov 3. PMID 30533549
- [Result] Harris-Love MO, Avila NA, Adams B, Zhou J, Seamon B, Ismail C, Zaidi SH, Kassner CA, Liu F, Blackman MR. The Comparative Associations of Ultrasound and Computed Tomography Estimates of Muscle Quality with Physical Performance and Metabolic Parameters in Older Men. J Clin Med. 2018 Oct 10;7(10):340. doi: 10.3390/jcm7100340. PMID 30308959